CLINICAL TRIAL: NCT01372722
Title: Phase I Study of Bilateral DBS to the Nucleus Accumbens (NAcc-DBS) for Treatment Resistant Bipolar Disorder
Brief Title: Deep Brain Stimulation (DBS) for Treatment Resistant Bipolar Disorder
Acronym: DBS-BIPO
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Other stimulation target (slMFB) more efficacious, unethical to continue with Nucleus Accumbens
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, MD, Professor of Psychiatry and Psychotherapy, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BSG-11-4712DBS
Record Dates: First submitted 2011-05-06; First posted 2011-06-14 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder
Keywords: treatment resistant
MeSH Terms: conditions — Bipolar Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham then Stimulation (Experimental)
  Interventions: Device: DBS Activa PC systems Medtronic
- Stimulation then Sham (Experimental)
  Interventions: Device: DBS, Activa PC systems Medtronic

INTERVENTIONS:
Device: DBS Activa PC systems Medtronic — 130Hz, 90us pulsewidth, 4V Amplitude
  Arms: Sham then Stimulation
Device: DBS, Activa PC systems Medtronic — 30Hz, 90us pulsewidth, 4V Amplitude
  Arms: Stimulation then Sham

SUMMARY:
Hypothesis to be tested:

Bilateral Deep Brain Stimulation to the Nucleus Accumbens is associated with clinically and statistically significant improvement in patients with treatment resistant bipolar disorder.

Overall Objective:

The aim in this interdisciplinary, psychiatric-neurosurgical project is to evaluate safety and efficacy of bilateral Deep Brain Stimulation to the Nucleus Accumbens (NAcc) using the Medtronic Activa RC Neurostimulator in patients with treatment resistant Bipolar Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years old. • German mother tongue • Ability to provide written informed consent.
* At least one manic or hypomanic episode according to DSM IV previous to onset of last depressive episode.
* Global Assessment of Function (GAF) score of > 46 • 5 years after the first episode of MD • DSM IV criteria for a current Major Depressive Episode (MDE) diagnosed by structured clinical interview for DSM IV. Diagnosis will be confirmed by two independent psychiatrists. • Current episode of MD > two years duration OR a history of more than 4 lifetime depressive episodes. • Minimum score at study entry of 28 on the 24-item Hamilton Depression Rating Scale (HDRS24).
* Average pre-operative HDRS24 score of 28 or greater (averaged over screening period) and a final preoperative HDRS24 score no more than 30% lower than the baseline screening HDRS score. • Treatment-resistant depression defined as: • Failure to respond to a minimum of four different antidepressant treatments, including medications and evidence-based psychotherapy (> 20 sessions with an experienced psychotherapist) administered at adequate doses and duration during the current episode. We will require documentation (i.e., statement from the treating psychiatrist) that a treatment trial has failed (either no response to maximum tolerable doses for a minimum of 5 weeks, or side-effects at sub-maximal doses) as coded by the Antidepressant Treatment History Form (ATHF). The study investigators will document each treatment by way of review of records from referring psychiatrists. • Failure or intolerance of an adequate course of electroconvulsive therapy (ECT) during any episode (> 6 bilateral treatments).
* A patient may remain on psychotropic medications during this study. However, doses must remain stable during a one month pre-operative evaluation period, the single blind phase and the open stimulation phase.

-If currently in psychotherapy, a patient must have been in this therapy for at least six months and continue to attend scheduled visits at no greater or lesser frequency than during the last three months. -

* Patients must have an established outpatient psychiatrist.
* Patients are able to fulfill the study requirements.
* Patients are in good general health.

Exclusion Criteria:

* Inability to tolerate general anesthesia.
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI)
* Cerebrovascular risk factors or a previous stroke, documented head trauma or neurodegenerative disorders.
* Other clinically significant Axis I psychiatric diagnoses including schizophrenia, bipolar I disorder (patients with bipolar II disorder will be included), panic disorder, obsessive-compulsive disorder, generalized anxiety disorder or post-traumatic stress disorder in the previous 12 months. Patients with severe Axis II personality disorders will also be excluded if they have the potential to interfere with cooperation during the pre- and post-operative phases of the study.
* Current psychotic symptoms.
* Current mixed episode.
* Evidence of global cognitive impairment.
* Substance abuse or dependence within the last year (except nicotine).
* Active suicidal ideation.
* Pregnancy and women of childbearing age not using effective contraception or currently nursing.
* General contraindications for DBS surgery (impossibility to conduct pre-operative fMRI, infections, claustrophobia, pregnancy, impossibility to stay awake during electrode implantation, medical risks regarding the operation, cardiac pacemaker/defibrillator or other implanted devices).
* Inability or unwillingness to comply with long-term follow-up.
* Patients who are not able to read and understand the consent form, or who are not capable of understanding or giving informed consent to the procedures of the study.
* History of intolerance to stimulation of any area of the body
* Participation in another drug, device or biologics trial within the preceding 30 days.
* Conditions requiring repeated MRI scans
* Conditions requiring diathermy
* Conditions requiring anticoagulant medication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Depression Severity rated with Montgomery Asberg Depression Scale (MADRS) | 12 month after DBS stimulation onset
  The Montgomery-Åsberg Depression Rating Scale (abbreviated MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. It was designed in 1979 by British and Swedish researchers as an adjunct to the Hamilton Rating Scale for Depression (HAMD) which would be more sensitive to the changes brought on by antidepressants and other forms of treatment than the Hamilton Scale is.
Young Mania Rating Scale (YMRS) | 12 month after DBS stimulation onset
  One of the most frequently used rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. This scale will be used to assess the development of manic symptoms over time, mainly in order to assess treatment emergent manic symptoms.

SECONDARY OUTCOMES:
Depression Severity rated with Hamilton Depression Rating Scale (HDRS24) | 12 month after DBS stimulation onset
  The Hamilton Rating Scale for Depression (HRSD), also known as the Hamilton Depression Rating Scale (HDRS) or abbreviated to HAM-D, is a multiple choice questionnaire that clinicians may use to rate the severity of a patient's major depression. The questionnaire rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. The questionnaire is presently one of the most commonly used scales for rating depression in medical research.
Adverse Event Schedule | 12 month after DBS stimulation onset
  Adverse events induced by the Stimulation will be recorded during the study using a structured questionnaire. 12 months after stimulation onset results will be compiled and rated as being due to DBS or not.
Comprehensive neuropsychological test battery | 12 month after DBS stimulation onset
  * General cognitive functions (Mini-Mental State Examination)
  * Attention (d2 attention-burden test)
  * Learning and memory tests covering verbal and visual spatial learning, memory and working memory (Verbal Learning and Memory Test, Rey Visual Design Learning Test,Wechsler Memory Scale)
  * language (HAWIE lexis tests, HAWIE finding similarities)
  * Executive functions (Trail Making Tests, Five-Point Test, and the Stroop test)
  * Visual perception (Hooper Visual Organization Test)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy - University Hospital, Bonn, Germany